CLINICAL TRIAL: NCT07092059
Title: Decentralized Clinical Trial of Contingency Management Digital Therapeutic to Treat Stimulant Use Disorder
Brief Title: Smartphone Services for Stimulant Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DynamiCare Health (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DCH003-StUD; R44DA059519 (NIH)
Record Dates: First submitted 2025-07-20; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Stimulant Use Disorder
Keywords: cocaine addiction; crack addiction; methamphetamine addiction; cocaine; crack; methamphetamine; stimulants; drug problem; drug addiction; drug abuse
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: This is a randomized control trial of a digital therapeutic.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- DynamiCare Group (Experimental): The main thing participants will do is use an app on their smartphone that might help with recovery. The most important feature of the app is that it allows participants to take a video selfie of themselves taking saliva (spit) drug tests. Then, the app will send these videos to the investigators in a way that is secure and protected. The app also has self-assessments & reading materials that may be of interest to participants. The intervention group will have an appointment and call tracking module and self-guided CBT therapy modules. The DynamiCare group will be able to report the data collected to their providers and will be able to share the app with people who support them.
  Interventions: Device: Smartphone digital therapeutic system
- Health & Wellness Group (Sham Comparator): The main thing participants will do is use an app on their smartphone that might help with their recovery. The most important feature of the app is that it allows participants to take a video selfie of themselves taking saliva (spit) drug tests. Then, the app will send these videos to the investigators in a way that is secure and protected. The app also has self-assessments & reading materials or modules that may be of interest to participants. The control group will have health and wellness information modules.
  Interventions: Device: Smartphone digital therapeutic system

INTERVENTIONS:
Device: Smartphone digital therapeutic system — This intervention is composed of a smartphone app (Apple iOS or Android type) that prompts patients with Stimulant Use Disorder to (1) complete self-assessment questionnaires in the app about their health, health care needs and the services they receive and other health-related functions in life, (2) read educational modules about health and wellness and answer questions about these readings, (3) speak periodically with a Guide about their use of the app, and (4) take periodic saliva substance tests using video-selfies with their smartphone camera. The intervention includes testing and interviews with the study staff over a 12 month period. There is a follow-up period to measure the longer-term results at 15 months, as well.

SUMMARY:
This study is testing two approaches to treating Stimulant Use Disorder, or problems with cocaine, crack, methamphetamine, etc. Stimulant Use Disorder is a national epidemic in the U.S. but there is no FDA-approved medication to treat it. There is a behavioral approach that has been found to be the most effective treatment for Stimulant Use Disorder, but this study is testing whether this can be delivered by a smartphone service, remotely, such as at home.

DETAILED DESCRIPTION:
We are trying to find out whether one version of a smartphone app is better than another in helping people who have stimulant use disorder. You will not be able to choose which app or app-based services you receive. You will be assigned to one of these two sets of smartphone-based services randomly - like by a flip of a coin. You have a 50/50 chance of receiving either version of the app.

You will need to agree to let us speak with your healthcare provider so that we can check this information about you before you start the study. We will also ask you to give us permission to look at how you use your health insurance. We want to learn if you are having visits to a clinic, doctors, Emergency Rooms, or hospitals. This is to learn if people get better and then use fewer healthcare services. We will check this information four times during the study. We will be able to see what treatments you have used, but we won't tell your insurance company that you are in this study. Also, we won't charge anything to your insurance.

ELIGIBILITY:
Inclusion Criteria:

* Adults who are at least 18 years old, speak/read English, have a smartphone, and who meet criteria for Stimulant Use Disorder, active or early remission. If being discharged to outpatient or intensive outpatient care, the patient is eligible.

Exclusion Criteria:

* Unwilling to authorize communication with any treatment provider(s), requiring acute detoxification from alcohol or opioids or residential or hospital treatment, or other obstacle to longitudinal participation in the study.
* Currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Saliva drug test outcomes | Testing will occur over a 15 month period.
  We will measure if your saliva drug tests show any use of drugs.

SECONDARY OUTCOMES:
Health outcomes | Assessments will occur over a 15 month period.
  We will ask you whether or not you are in treatment, whatever healthcare services you use (such as Emergency Room visits, hospital stays), the ways in which you use the app, and about your health and other health functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Carla J Rash, PhD, Principal Investigator — UConn Health; David R Gastfriend, MD, Principal Investigator — DynamiCare Health Inc.
Locations (1):
- This is an At-Home Study - no travel or on-site visits are needed at all; Main Office: 6 Liberty Sq, #2102, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided